CLINICAL TRIAL: NCT01637207
Title: How Easy is it to Identify the Cricothyroid Membrane in Children? Can Ultrasound Imaging me Used to Aid Identification?
Brief Title: How Easy is it to Identify the Cricothyroid Membrane in Children? Can Ultrasound Imagine be Used to Aid Identification?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10AR11
Record Dates: First submitted 2012-06-01; First posted 2012-07-11 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Cricothyroidotomy
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- palpation (Experimental)
  Interventions: Other: Palpation
- ultrasound (Experimental)
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Palpation — Group A: Palpation Group
  Arms: palpation
Other: Ultrasound — Group B: Ultrasound Group
  Arms: ultrasound

SUMMARY:
The Investigators aim to determine how easy it is for anaesthetists to identify the Cricothyroid membrane (CTM) in children and infants and whether ultrasound maybe useful in addition. The investigators aim to conduct a randomised single blinded trial to compare methods to detect the CTM.

The first group of patients will be randomised to palpation of anatomical landmarks group. Prior to commencing the MRI scan the anaesthetist is timed to identify the CTM and then the trachea using a felt tip pen. A ficidual marker will be placed on the 2 marked areas.

The second group of patients will be randomised to receive ultrasound. Prior to commencing the MRI scan the sonographer is timed to identify the CTM and then the trachea using a felt tip pen. A ficidual marker will be placed on the two marked areas.

DETAILED DESCRIPTION:
Cricothyroidotomy is an infrequent but potentially life-saving procedure. The need for cricothyroidotomy arises from the can't intubate and can't ventilate (CICV) scenario and is therefore incorporated in the difficult airway guidelines for both adults and children. This CICV scenario is less common in the paediatric population than in the adult population and most difficult airways can be managed with-bag mask ventilation and PEEP.

The cricothyroid membrane is a useful place to access the airway in the case of glottic or supraglottic obstruction as it is relatively avascular, superficial and the 'full ring' of the cricoid protects against posterior perforation. In adults, the average the cricothyroid membrane CTM is 13.7mm long and 12.4mm wide. The CTM is relatively short in children. In neonates the CTM has a mean height of 2.6mm and a width of 3mm.

In children the most prominent anterior midline structures in the neck are not the thyroid as in adults but the hyoid bone and cricoid cartilage. As the larynx is more cephalad in children the cricothyroid membrane is higher than in adults and placement of a catheter may be more difficult as the mandible gets in the way. A healthy amount of adipose in the subcutaneous tissue can obscure the anatomy. Currently clinicians identify the CTM using palpation of anatomical landmarks. In infants, with the head in extension and soft tissue pulled up towards the mandible, the CTM may be difficult to distinguish. It is suggested that bimanual manipulation may enable identification of the cartilaginous trachea.

To perform a cricothyroid puncture, a syringe containing sterile saline is attached to a cannula. The skin over the cricothyroid membrane is stabilised with the index finger and thumb of the non-dominant hand. The transtracheal cannula is inserted through the cricothyroid membrane at a 45º angle heading caudal and posterior. However, in neonates due to the restricted dimensions, a needle is the only option for cricothyroidotomy. Even in experienced hands, cricothyroidotomy is technically challenging. In inexperienced hands this can lead to significant injuries including the risk of fracture of the thyroid and cricoid cartilages.

A recent abstract has tried to determine whether how easy it is to locate the CTM in children. Their initial conclusions suggest that the identification of the CTM is difficult. The limitations of their study are that there are small numbers and only one person has been asked to perform the identification.

The applications of ultrasound are vast and varied. It is readily available, portable and easy to use. Of note, a recent study has used ultrasound (Sonosite 10Hz) to help identify the CTM in adults. Following a period of training, it was found to improve accuracy and speed of identification.

The investigators aim to determine how easy it is for anaesthetists to identify the CTM in children and infants and whether ultrasound maybe a useful adjunct. The investigators aim to conduct a randomized single blinded trial to compare methods to detect the CTM: palpation of anatomical landmarks versus ultrasound .

ELIGIBILITY:
Inclusion Criteria:

* All children between 0-8 years requiring general anaethesia for elective MRI head, neck and spinal scans

Exclusion Criteria:

* Children with obvious neck deformity, goitre, tracheostomy and emergency cases

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of placement of the marker | 4-6 months
  Accuracy of the placement of the marker in relation to the cricithyroid membrane and trachea on MRI images.

SECONDARY OUTCOMES:
Time taken to identify CTM/Trachea | 4-6 months
  Time taken to identify CTM/Trachea placement confidence assessed using the VAS Score (0-100: impossible to very confident). Comparison between age groups 0-4 years Vs 4-8 years.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Dobby, MBBS, Principal Investigator — Great Ormond Street Hospital for Sick Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Sick Children NHS Foundation Trust, London, United Kingdom